CLINICAL TRIAL: NCT04454047
Title: Extracapsular Arthroscopic Treatment for Refractory Tennis Elbow--Mid-and-short Term Retrospective Study of 50 Cases
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2017421
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Tennis Elbow
Keywords: Refractory tennis elbow; Arthroscopy; Intracapsular method; Extracapsular method; Surgical technology
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Extracapsular method group: 50 patients with refractory tennis elbow who received extracapsular arthroscopic surgery.
  Interventions: Procedure: Extracapsular arthroscopy

INTERVENTIONS:
Procedure: Extracapsular arthroscopy — Extracapsular arthroscopy method was used to treat refractory tennis elbow

SUMMARY:
This study retrospectively analysed surgical outcomes of consecutive 50 cases to investigate the technical standard and clinical effect of extracapsular arthroscopic treatment for refractory tennis elbow.

DETAILED DESCRIPTION:
To investigate the technical standard of extracapsular arthroscopic treatment for refractory tennis elbow. Consecutive 50 cases of refractory tennis elbow from 50 patients who underwent extracapsular arthroscopic surgery which performed independently by the same doctor from March 2012 to November 2016 was retrospectively analyzed. The key points of technical standard were summarized, including debridement, decortication and microfracture, suture under arthroscopy and postoperative cast fixation. Visual Analogue Scale(VAS), Mayo elbow performance score and Disability of Arm, Shoulder, and Hand outcome measure (DASH) were evaluated for postoperative results. The effects of various technical points were analyzed by rank sum test, independent sample t test, χ2 test and multiple logistic regression.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis was refractory tennis elbow;
2. Standard extracapsular method was used for surgery.

Exclusion Criteria:

1. Patient had past history of joint infection, joint tuberculosis, or osteomyelitis, or the upper limb had undergone surgery within the past 6 months;
2. Diagnosis was combined with severe heart, brain, kidney, or another organ dysfunction;
3. Case was complicated with other serious elbow joint diseases or injuries;
4. Patient did not sign the informed consent form.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The quantitative data of 50 patients (20 men and 30 women) were reviewed. The minimum age was 35 years, and the maximum age was 55 years old, with an average of 44.6 years.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Mayo Elbow Performance Score | 24 months
  Use Mayo Elbow Performance Score（MEPS） to evaluate the functional recovery of patients who received extracapsular arthroscopic treatment. MEPS ranges from 0 to 100, higher scores mean a better outcome.
Visual Analog Scale | 24 months
  Use Visual Analog Scale(VAS) to evaluate the pain recovery of patients who received extracapsular arthroscopic treatment. VAS ranges from 0 to 10, higher scores mean a worse outcome.
Disability of Arm, Shoulder and Hand score | 24 months
  Use Disability of Arm, Shoulder and Hand(DASH) score to evaluate the functional and pain recovery of patients who received extracapsular arthroscopic treatment. DASH ranges from 0 to 100, higher scores mean a worse outcome.
Activity of Daily Life recovery time | 24 months
  Use Activity of Daily Life(ADL) recovery time to evaluate the functional recovery of patients who received extracapsular arthroscopic treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Univerisity Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No